CLINICAL TRIAL: NCT00334880
Title: A Phase III, Randomized, Double-Blind, Multi-Center, Placebo-Controlled, Parallel-Group, Forced Dose Titration, Safety and Efficacy Study of NRP104 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study to Assess the Safety and Efficacy of NRP104 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NRP104.303
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders With Hyperactivity; Attention Deficit Hyperactivity Disorders
Keywords: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders with Hyperactivity; Attention Deficit Hyperactivity Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NRP104

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of NRP104 administered as a daily morning dose (30, 50, and 70mg/day) compared to placebo in adults (18-55 years of age inclusive) diagnosed with moderate to severe Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This study is a randomized, phase III, multi-center, placebo-controlled, parallel-group, forced dose titration in which adult subjects (18-55 years of age inclusive) with ADHD will be randomized to NRP104 (30, 50, or 70 mg) or placebo for four weeks of double-blind evaluation of safety and efficacy.

The study will have three phases: (1) screening and washout; (2) baseline; and (3) 4-week double-blind evaluation of NRP104 and placebo. The double-blind period will include a forced dose titration phase followed by a fixed dose phase. Subjects will be required to visit the site up to 6 times over a 5-8 week period, or longer in cases requiring a 28-day wash out.

Screening and Washout: Subjects will be screened to establish eligibility for study participation. The Screening Visit (Visit 1) may take place over multiple days if needed to accommodate the subject's schedule. Those subjects who meet eligibility requirements will undergo medication washout, if applicable. The length of the ADHD medication washout period will range from 7-28 days.

Baseline: Following medication washout, subjects will return to the clinic for reassessment of eligibility criteria and establishment of baseline measures. The interval between the first day of the Screening Visit (informed consent date) and the Baseline Visit (Visit 2) must not exceed 35 days. Eligible subjects with a baseline ADHD-RS score greater than or equal to 28 (performed using adult DSM-IV prompts) will be randomized to treatment.

Double-blind treatment: Eligible subjects will be randomly assigned (in a 2:2:2:1 ratio of each of the three active doses vs. placebo) to a daily morning dose of NRP104 or placebo for 4 weeks. All NRP104 groups will start at a dose of 30 mg/day. Subjects randomized to 70 mg will be titrated to that dose over a 2-week period; those randomized to 50 mg will be titrated to that dose over a 1-week period; and those randomized to 30 mg will begin dosing on 30 mg per day during week one and will remain on that dose throughout the study. Double-blind assessment of the safety and efficacy of NRP104 will proceed for 4 weeks with weekly clinic visits scheduled for evaluations and medication disbursement.

Follow-up period: Subjects who have completed at least 2 weeks of double-blind participation, will have the option to continue participation in an open-label extension study (Protocol NRP104.304: one-year safety study). Subjects who are not eligible or who choose not to participate in the extension study will continue to be followed for thirty days following their last dose of study drug. A telephone contact (or contact in person) will be initiated by the research site to collect any new or ongoing SAEs and to follow-up on any unresolved or related AEs from the Final Study Visit or Early Termination (ET) Visit (Visit 6). If the Principal Investigator determines AEs are not acceptably resolved, appropriate follow-up should continue until all safety concerns, in the opinion of the Investigator, are resolved.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18-55 years of age, inclusive.
* Must be male or non-pregnant female. Females of childbearing potential (FOCP) must use contraception.
* Must have a medical assessment with no clinically significant or relevant abnormalities as determined by medical history, PE, clinical and lab evaluation.
* Must have 12-lead ECGs defined by the following parameters:

  1. QT/QTcF interval < 450 msec for males and < 470 msec for females
  2. Resting heart rate is between 40 and 100 beats per minute
  3. P-R interval < 200 msec
  4. QRS interval <110 msec.
* Meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM-IV-TR™) criteria for a primary diagnosis of ADHD (diagnostic code 314.00 and 314.01) established by a psychiatric evaluation that reviews DSM-IV-TR™ criteria with at least 6 of the 9 subtype criteria met. The Adult ADHD Clinical Diagnostic Scale (ACDS v1.2) will be utilized as the diagnostic tool.
* Has a baseline ADHD-RS score greater than or equal to 28 assessed using adult DSM-IV prompts.
* Understands and is able, willing, and likely to fully comply with the study procedures and restrictions.
* Has given written informed consent to participate in the study in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines and applicable regulations before completing any study procedures.

Exclusion Criteria:

* In the opinion of the investigator, the subject is significantly underweight [e.g., Body Mass Index (BMI) < 18.5] or morbidly obese.
* Has any comorbid psychiatric diagnosis with significant symptoms such as any severe comorbid Axis II disorders or severe Axis I disorders including Post Traumatic Stress Disorder (PTSD), psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder or other symptomatic manifestations that will contraindicate NRP104 treatment or confound efficacy or safety assessments. Specifically, subjects with mild to moderate forms of Axis I disorders including social phobia and dysthymia may be included while subjects with a lifetime history of psychosis or bipolar disorder will be excluded from participation. Comorbid psychiatric diagnoses will be established by a psychiatric evaluation that includes the Structured Clinical Interview for DSM-IV-TR™ disorders (SCID-I) interview at the screening visit.
* Has any concurrent chronic or acute illness or unstable medical condition that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol. Subjects with mental retardation or a severe learning disability are excluded.
* Has a history of seizure (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
* Has a known cardiac structural abnormality or any other condition that may affect cardiac performance.
* Has any clinically significant ECG or laboratory abnormality at Screening or Baseline.
* Subject has a history of hypertension or has a resting sitting systolic blood pressure > 139mmHg or diastolic blood pressure > 89mmHg.
* Has used any prohibited medication except for ADHD medications within 30 days of screening visit. Hormonal contraceptives are acceptable.
* Has a documented allergy, intolerance, or documented history of non-responsivity to methylphenidate or amphetamine.
* Currently has (or had a history within the last 6 months of) a drug dependence or substance abuse disorder according to DSM-IV-TR™ criteria (excluding nicotine) as established by a SCID-I at the screening visit.
* Has a positive urine drug result at Screening (with the exception of subject's current stimulant therapy, if any) or at Baseline.
* Has taken an investigational drug or taken part in a clinical trial within 30 days prior to Screening.
* The female subject is pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2006-05; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Clinician-administered ADHD-rating scale (ADHD-RS) performed using adult DSM-IV prompts | weekly over a period of 4 weeks

SECONDARY OUTCOMES:
The Clinical Global Impression of Improvement (CGI-I) | 4 times over a period of 4 weeks
Self-report of the Pittsburgh Sleep Quality Index (PSQI) measured at Baseline and at the Final Study Visit | twice over a period of 4 weeks
Occurrence of treatment-emergent adverse events and specific evaluation of blood pressure, heart rate, electrocardiogram (ECG), laboratory findings, and physical examination (PE) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (48):
- United States (48):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - University of California, Irvine Child Development Center, Irvine, California
  - Bay Area Research Institute, Lafayette, California
  - Peninsula Research Associates, Rolling Hills Estate, California
  - University of California, San Francisco, Dept. of Psychiatry, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Psychiatric Medicine Center, New London, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Janus Center for Psychiatric Research LLC, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Carman Research, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Johns Hopkins at Green Spring Station, Lutherville, Maryland
  - Marc Hertzman, MD, Rockville, Maryland
  - Massachusetts General Hospital, Cambridge, Massachusetts
  - Summit Research Network (Michigan) Inc., Flint, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - St Charles Psychiatric Associates-Midwest Research, Saint Charles, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - CNS Research Institute (CRI), Clementon, New Jersey
  - VA NY Harbor Healthcare System, New York, New York
  - Duke University ADHD Program, Durham, North Carolina
  - Richard Weisler and Associates, Raleigh, North Carolina
  - University Hospitals of Cleveland, Case Western Reserve University, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - CNS Research Institute, P.C., Philadelphia, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - Bayou City Research, Houston, Texas
  - Red Oak Psychiatry Associates, P.A., Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - John M. Turnbow, MD, PA, Lubbock, Texas
  - The Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Psychiatric Alliance of the Blue Ridge Clinical Research, Charlottesville, Virginia
  - NeuroScience, Inc., Herndon, Virginia
  - Brighton Research Group, Virginia Beach, Virginia
  - Summit Research Network LLC (Seattle), Seattle, Washington

REFERENCES:
- [Result] Adler LA, Goodman DW, Kollins SH, Weisler RH, Krishnan S, Zhang Y, Biederman J; 303 Study Group. Double-blind, placebo-controlled study of the efficacy and safety of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2008 Sep;69(9):1364-73. doi: 10.4088/jcp.v69n0903. Epub 2008 Sep 9. PMID 19012818
- [Derived] Schein J, Cloutier M, Gauthier-Loiselle M, Catillon M, Xu C, Chan D, Childress A. Assessment of centanafadine in adults with attention-deficit/hyperactivity disorder: A matching-adjusted indirect comparison vs lisdexamfetamine dimesylate, atomoxetine hydrochloride, and viloxazine extended-release. J Manag Care Spec Pharm. 2024 Jun;30(6):528-540. doi: 10.18553/jmcp.2024.30.6.528. PMID 38824626
- [Derived] Mattingly GW, Weisler RH, Young J, Adeyi B, Dirks B, Babcock T, Lasser R, Scheckner B, Goodman DW. Clinical response and symptomatic remission in short- and long-term trials of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder. BMC Psychiatry. 2013 Jan 29;13:39. doi: 10.1186/1471-244X-13-39. PMID 23356790
- [Derived] Babcock T, Dirks B, Adeyi B, Scheckner B. Efficacy of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder previously treated with amphetamines: analyses from a randomized, double-blind, multicenter, placebo-controlled titration study. BMC Pharmacol Toxicol. 2012 Dec 19;13:18. doi: 10.1186/2050-6511-13-18. PMID 23254273
- [Derived] Surman CB, Roth T. Impact of stimulant pharmacotherapy on sleep quality: post hoc analyses of 2 large, double-blind, randomized, placebo-controlled trials. J Clin Psychiatry. 2011 Jul;72(7):903-8. doi: 10.4088/JCP.11m06838. PMID 21824454
- [Derived] Waxmonsky JG, Waschbusch DA, Glatt SJ, Faraone SV. Prediction of placebo response in 2 clinical trials of lisdexamfetamine dimesylate for the treatment of ADHD. J Clin Psychiatry. 2011 Oct;72(10):1366-75. doi: 10.4088/JCP.10m05979pur. PMID 21367347
- [Derived] Adler LA, Weisler RH, Goodman DW, Hamdani M, Niebler GE. Short-term effects of lisdexamfetamine dimesylate on cardiovascular parameters in a 4-week clinical trial in adults with attention-deficit/hyperactivity disorder. J Clin Psychiatry. 2009 Dec;70(12):1652-61. doi: 10.4088/JCP.09m05335pur. PMID 20141706
- [Derived] Adler LA, Goodman D, Weisler R, Hamdani M, Roth T. Effect of lisdexamfetamine dimesylate on sleep in adults with attention-deficit/hyperactivity disorder. Behav Brain Funct. 2009 Aug 3;5:34. doi: 10.1186/1744-9081-5-34. PMID 19650932
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html